CLINICAL TRIAL: NCT01855737
Title: Clinical Study of the Relationship Between Pharmacogenomics and Warfarin Dose in Chinese Patients
Brief Title: The Study of Warfarin Maintenance Dose in Chinese Patients
Acronym: WADCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Hong Liu, Key Laboratory of Clinical Trial Research in Cardiovascular Drugs, Ministry of Health, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2011-GZH1
Record Dates: First submitted 2013-05-06; First posted 2013-05-16 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Atrial Fibrillation; Heart Valve Disease; Pulmonary Artery Embolism
Keywords: gene guided; warfarin dose; Chinese
MeSH Terms: conditions — Atrial Fibrillation; Heart Valve Diseases; Pulmonary Embolism | interventions — Warfarin

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA frozen in -80℃
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Warfarin Using Group
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Prescribe warfarin to the patients who are needed.
  Other Names: Manufacturer: Orion Corporation; Product Name: Warfarin; 3mg*100

SUMMARY:
1. Title: Clinical study of the relationship between Pharmacogenomics and warfarin dose in Chinese patients
2. Drug: Warfarin
3. Design: To value the accuracy of warfarin Pharmacogenomics algorithm by the algorithm calculated dose and actual dose in the Chinese patients.
4. Hypothesis:Pharmacogenomic algorithm guided dose can help to predict warfarin dose in Chinese patients.

DETAILED DESCRIPTION:
* For the patients who need to use warfarin, detect the "Vitamin K epoxide reductase complex subunit 1 (VKORC1),cytochrome p450 2C9 (CYP2C9), and cytochrome p450 4F2 (CYP4F2) genotype.
* Record the demographic information: gender, age, height, and weight.
* Record drug combination, complications, and international normalized ratio (INR), liver function and kidney function or other biochemical test results.
* Put genotypes, demographic information and other clinical information into the algorithm to calculate warfarin dose for the patients, and compared with the actual dose.

ELIGIBILITY:
Inclusion Criteria:

* Chinese patients
* Age >18y
* target INR 1.5~3.0
* Patients signed informed consent

Exclusion Criteria:

* Has hemorrhage disease, or tendency to significant bleeding
* Severe liver and kidney disfunction, serious infections, severe heart failure (NYHA heart function classification Ⅲ magnitude), severe pulmonary hypertension, abnormal thyroid function, respiratory failure, anemia, malignant tumor, blood disease
* patients with pregnancy or lactation;
* with cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Han population who need to use Warfarin and older than 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the pharmacogenomics algorithm for warfarin maintenance dose | one month after the initial dose of warfarin
  The proportion of the patients whose predicted dose were within 20% of the actual maintenance dose.

CONTACTS AND LOCATIONS:
Overall Officials: Yishi Li, MD, PhD, Principal Investigator — Key Laboratory of Clinical Trial Research in Cardiovascular Drugs, Ministry of Health, Cardiovascular Institute and Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College; Hong Liu, MS, Principal Investigator — Key Laboratory of Clinical Trial Research in Cardiovascular Drugs, Ministry of Health, Cardiovascular Institute and Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Key Laboratory of Clinical Trial Research in Cardiovascular Drugs, Ministry of Health, Cardiovascular Institute and Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China